CLINICAL TRIAL: NCT03451825
Title: Open-label, Phase I/II Study to Evaluate Pharmacokinetics, Pharmacodynamics, Safety, and Anticancer Activity of Avelumab in Pediatric Subjects From Birth to Less Than 18 Years of Age With Refractory or Relapsed Solid Tumors and Lymphoma
Brief Title: Phase I/II Study of Avelumab in Pediatric Cancer Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the limited activity observed with avelumab monotherapy in the pediatric population, the Phase II study part was cancelled.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS100070-0306; 2017-002985-28 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Refractory or Relapsed Solid Tumors; Lymphoma
Keywords: Avelumab; Anti PD-L1; Solid tumors; CNS tumors; Lymphoma; Pediatric subjects
MeSH Terms: conditions — Lymphoma; Central Nervous System Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avelumab: 10 miligram per kilogram (mg/kg) (Experimental)
  Interventions: Drug: Avelumab
- Avelumab 20mg/kg (Experimental)
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Participants received an intravenous infusion of avelumab 10mg/kg intervention (IV) once every 2 weeks until confirmed progression, death, unacceptable toxicity, or any criterion for withdrawal occurred.
  Arms: Avelumab: 10 miligram per kilogram (mg/kg)
Drug: Avelumab — Participants received an intravenous infusion of avelumab 20mg/kg intervention (IV) once every 2 weeks until confirmed progression, death, unacceptable toxicity, or any criterion for withdrawal occurred.
  Arms: Avelumab 20mg/kg

SUMMARY:
This is a multi-center, open-label, international study to evaluate the dose, safety and tolerability, antitumor activity, pharmacokinetic and pharmacodynamics of avelumab in pediatric subjects 0 to less than 18 years of age with refractory or relapsed malignant solid tumors (including central nervous system tumors) and lymphoma for which no standard therapy is available or for which the subject is not eligible for the existing therapy.

The study was planned to be conducted in 2 parts: the dose-finding part (Phase I) and the tumor-specified expansion part (Phase II). However, Phase II was cancelled due to limited clinical benefit of PD-L1 monotherapy in pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 0 to less than 18 years of age at the time of first treatment dose with histologically or cytologically confirmed solid malignant tumors (including CNS tumors) or lymphoma for which no standard therapy is available
* Confirmed progression on or refractory to standard therapy or no standard therapy available.
* Availability of archival formalin-fixed, paraffin-embedded block containing tumor tissue, or slides, or a fresh/recent tumor biopsy prior to avelumab treatment for subjects in Phase 2
* Adequate bone marrow, kidney, and liver function
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Prior therapy with any antibody or drug targeting T-cell coregulatory proteins
* Concurrent anticancer treatment or immunosuppressive agents
* Prior organ transplantation
* Significant acute or chronic infections
* Other significant diseases or conditions that might impair the subject's tolerance of trial treatment
* Other protocol defined exclusion criteria could apply

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (11):
- United States (2):
  - Children's Hospital Colorado, Aurora, Colorado
  - The Children's Hospital at Montefiore (CHAM), The Bronx, New York
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Leuven, Leuven
- Canada (3):
  - Children's Hospital - London Health Sciences Centre, London
  - CHU Sainte-Justine, Montreal
  - The Hospital for Sick Children, Toronto
- Rigshospitalet, Copenhagen, Denmark
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul

REFERENCES:
- [Result] Vugmeyster Y, Grisic AM, Brockhaus B, Rueckert P, Ruisi M, Dai H, Khandelwal A. Avelumab Dose Selection for Clinical Studies in Pediatric Patients with Solid Tumors. Clin Pharmacokinet. 2022 Jul;61(7):985-995. doi: 10.1007/s40262-022-01111-8. Epub 2022 Apr 29. PMID 35484319
- [Result] Loeb DM, Lee JW, Morgenstern DA, Samson Y, Uyttebroeck A, Lyu CJ, Van Damme A, Nysom K, Macy ME, Zorzi AP, Xiong J, Pollert P, Joerg I, Vugmeyster Y, Ruisi M, Kang HJ. Avelumab in paediatric patients with refractory or relapsed solid tumours: dose-escalation results from an open-label, single-arm, phase 1/2 trial. Cancer Immunol Immunother. 2022 Oct;71(10):2485-2495. doi: 10.1007/s00262-022-03159-8. Epub 2022 Mar 9. PMID 35262780
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070-0306
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 26 participants were screened for participation in the Phase I part of the study, out of which 21 participants were eligible and received the study treatment.
Pre-assignment Details: The study was planned to be conducted in 2 parts: the dose-finding part (Phase I) and the tumor-specified expansion part (Phase II). However, Phase II was cancelled due to limited clinical benefit of Programmed death ligand 1 (PD-L1) monotherapy in pediatric participants.
Groups:
- Avelumab 10 Miligram Per Kilogram (mg/kg): Participants received an intravenous infusion of avelumab 10mg/kg intervention (IV) once every 2 weeks until confirmed progression, death, unacceptable toxicity, or any criterion for withdrawal occurred.
- Avelumab 20 mg/kg: Participants received an intravenous infusion of avelumab 20 mg/kg IV once every 2 weeks until confirmed progression, death, unacceptable toxicity, or any criterion for withdrawal occurred.
Period: Overall Study
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Started | 6 | 15
Completed | 6 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who had received any dose of avelumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg | Total
Number analyzed (Participants) | 6 | 15 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.0 (3.10) | 10.7 (5.02) | 11.1 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 10
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 13 | 19
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 4 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) as Per Severity With Grade 3 or Higher According to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 4.03 (NCI-CTCAE v4.03)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant, which does not necessarily have causal relationship with treatment. A serious AE was defined as an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged in participant hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were those events with onset dates occurring during the on-treatment period for the first time, or if the worsening of an event was during the on-treatment period. TEAEs included both serious TEAEs and non-serious TEAEs. Severity of grade 3 or higher TEAEs were graded using NCI-CTCAE v4.03 toxicity grades, as follows: Grade 1 = Mild, Grade 2= Moderate, Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with TEAEs as per severity with Grade 3 and higher were reported.
Time Frame: Baseline up to 1182 days
Population: Safety analysis set included all participants who received any dose of avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants
  Participants With TEAEs: Grade 3 | 4 | 6
  Participants With TEAEs: Grade 4 | 0 | 2
  Participants With TEAEs: Grade 5 | 1 | 3

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: For the purpose of dose finding, any of the following AEs occurring during the primary DLT observation period. Hematologic: Grade 4 neutropenia for more than 7 days in duration; Grade greater than or equal to (>=) 3 neutropenic infection; Grade >= 3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia > 7 days and Grade 4 anemia. Nonhematologic: Any Grade >= 3 toxicity, except for any of the following: Transient (less than or equal to (<=) 72 hours; Grade 3 flu-like symptoms or fever, which was controlled with medical management; Transient (<= 72 hours) Grade 3 fatigue, local reactions, headache, nausea, or emesis that resolved to Grade <= 1 or to Baseline. Grade 3 diarrhea or Grade 3 skin toxicity that resolved to Grade <= 1 in less than 7 days after medical management (immunosuppressant treatment) had been initiated. Grade >= 3 amylase or lipase abnormality that was not associated with clinical manifestations of pancreatitis.
Time Frame: Baseline up to 28 days
Population: The DLT analysis set includes all participants who meet either of the following criteria: Have received 100 percent (% ) of all planned doses of treatment during the DLT evaluation period (first 2 cycles of treatment) and have been followed for at least 28 days or have stopped treatment because of a DLT in the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 12
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With Confirmed Best Overall Response (BOR) as Per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) and as Adjudicated by the Investigator
Description: Confirmed BOR was evaluated based on RECIST v1.1 and Investigator's assessments and defined as best response of any of confirmed complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) recorded from date of study treatment until disease progression. CR: Disappearance of all evidence of target/non-target lesions. PR: At least 30 percent (%) reduction from baseline in sum of longest diameter (SLD) of all lesions. SD: Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD: at least a 20% increase in SLD, taking as reference smallest SLD recorded from baseline/appearance of 1or more new lesions and unequivocal progression of non-target lesions.
Time Frame: Baseline up to 1182 days
Population: Full analysis set included all participants who received any dose of avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Stable Disease (SD) | 0 | 4
  Non-CR/Non-PR | 0 | 0
  Progressive Disease (PD) | 5 | 9
  Not Evaluable | 1 | 2

4. Secondary Outcome: Duration of Response (DOR) as Per Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) and as Adjudicated by the Investigator
Description: Duration of response was defined for participants with confirmed objective response (OR), as the time from first documentation of objective response (Complete Response or Partial Response) to the date of first documentation of objective PD or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. DOR was determined according to RECIST v1.1 and assessed by Investigator.
Time Frame: Time from first documentation of objective response up to 1182 days
Population: Data could not be calculated as none of the participants showed objective response.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Response According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) and as Adjudicated by the Investigator
Description: Time to response (TTR) was defined, for participants with an objective response, as the time from the start date of study treatment to the first documentation of OR (CR or PR) which was subsequently confirmed.
Time Frame: Time from start of study treatment up to 1182 days
Population: Data could not be calculated as none of the participants showed confirmed objective response.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression-Free Survival According to Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1) and as Adjudicated by the Investigator
Description: Progression-Free survival was defined as the time from first administration of study treatment until the first documentation of disease progression (PD) or death due to any cause, whichever occurred first. PD: At least a 20 % increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from first administration of study drug until the first documentation of PD or death, assessed up to 1182 days
Population: Full analysis set included all participants who received any dose of avelumab. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 12
Weeks | 7.5 (6.57) [6.57 to 8.14] | 7.7 (0.14) [0.14 to 131.86]

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as the time from date of first dose of study drug to the date of death due to any cause. For participants who were still alive at the time of data analysis or who were lost to follow-up, OS time was censored at the date of last contact. OS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Time from first administration of study drug up to 1182 days
Population: as for outcome 6
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 12
Months | 4.4 (1.51) [1.51 to 14.36] | 7.0 (0.85) [0.85 to 31.97]

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events, Adverse Events of Special Interest (AESI) and Treatment-related Adverse Events According to NCI-CTCAE v4.03
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs was defined as events with onset date or worsening during the on-treatment period. TEAEs included serious AEs and non-serious AEs. Treatment-related TEAEs: reasonably related to the study intervention. AESIs included Infusion-related reactions (IRRs) and Immune-related AE (irAEs).
Time Frame: Baseline up to 1182 days
Population: The safety analysis set included all participants who received any dose of avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants
  Participants with any TEAEs | 6 | 15
  Participants with Treatment-emergent irAE | 0 | 1
  Participants with Treatment-emergent IRR | 2 | 7
  Participants with Study-drug related TEAEs | 3 | 10

9. Secondary Outcome: Number of Participants With Grade 3 or Higher Laboratory Abnormalities According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03
Description: The total number of participants with laboratory test abnormalities were assessed. Clinical laboratory tests included hematology and biochemistry abnormalities. The hematology and biochemistry abnormalities (by worst on-treatment NCI-CTCAE Grade 3 and Grade 4) were reported. Laboratory abnormalities were graded using NCI-CTCAE v4.03 toxicity grades, as follows: Grade 1 = Mild, Grade 2= Moderate, Grade 3 = Severe; Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: Baseline up to 1182 days
Population: Safety analysis set included all participants who received any dose of avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants
  Grade 3: Anemia: | 1 | 1
  Grade 3: lymphocyte count decreased | 1 | 2
  Grade 4: platelet count decreased | 0 | 1
  Grade 3: hyponatremia | 1 | 3
  Grade 3: hyperkalemia | 1 | 0
  Grade 3: creatinine increased | 1 | 0
  Grade 3: alkaline phosphatase increased | 1 | 1
  Grade 3: hypokalemia | 0 | 2
  Grade 3: serum amylase increased | 0 | 1
  Grade 4: Hyperkalemia | 0 | 1

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Avelumab
Description: Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, end of infusion (1 hour), 3 hours post-dose on Day 1, cycle 1 (each cycle is for 14 days)
Population: The Pharmacokinetic (PK) analysis set included all participants who received at least one dose of avelumab, had no important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per mililiter (mcg/mL)
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
microgram per mililiter (mcg/mL) | 190 (34.5) [lower limit 34.5] | 384 (27.3) [lower limit 27.3]

11. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to the 336 Hours Post-Dose (AUC 0-336 Hours) of Avelumab
Description: Area under the serum concentration-time curve from time zero to the 336 Hours Post-Dose (AUC 0-336 hours) of Avelumab were calculated. Calculated using the mixed loglinear trapezoidal rule (linear up, log down).
Time Frame: Pre-dose, end of infusion (1 hour), 3 hours to 336 hours post-dose
Population: The PK analysis set included all particpants who received at least one dose of avelumab, had no important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration. Here" number of participants analyzed" are those who are evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per mililiter (mcg•h/mL)
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 14
microgram*hour per mililiter (mcg•h/mL) | 18800 (29.2) [lower limit 29.2] | 43500 (21.5) [lower limit 21.5]

12. Secondary Outcome: Apparent Terminal Half Life (t1/2) of Avelumab
Description: Apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination. Apparent terminal half-life. t1/2 = log (ln) 2/lambdaz (λz).
Time Frame: Pre-dose, end of infusion (1 hour), 3 hours post-dose on Day 1, cycle 1 (each cycle is for 14 days)
Population: The PK analysis set included all participants who received at least one dose of avelumab, had no important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration. Here, "Number of participants analyzed" are those who are evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 4 | 7
hours | 85.9 (15.1) [15.1 to 102] | 119 (73.7) [73.7 to 486]

13. Secondary Outcome: Minimum Serum Post-dose Trough (Ctrough) Concentration of Avelumab
Description: The concentration observed immediately before next dosing (corresponding to predose or trough concentration for multiple dosing) was calculated.
Time Frame: Pre-dose at Day 15
Population: The PK analysis set included all participants who received at least one dose of avelumab, had no important protocol deviations or important events affecting PK, and provided at least one measurable post-dose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per ml (mcg/mL)
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 14
microgram per ml (mcg/mL) | 11.2 (44.9) [lower limit 44.9] | 34.8 (77.8) [lower limit 77.8]

14. Secondary Outcome: Number of Participants With Positive Treatment Emergent Anti-drug Antibodies (ADA) and Neutralizing Antibodies (Nabs)
Description: Serum samples were analyzed by a validated electrochemiluminesce immunoassay to detect the presence of anti-drug antibodies and neutralizing antibodies. Samples that screened positive were subsequently tested in a confirmatory assay. Those confirmed positive were tittered for a quasi-quantitative result. Number of participants with positive treatment emergent anti-drug antibodies and neutralizing antibodies were reported. Participants not positive prior to treatment with avelumab and with at least one positive result in the human-Antihuman Antibodies assay were characterized as treatment-emergent.
Time Frame: Baseline up to 1182 days
Population: Immunogenicity Analysis Set included all partiicpants who received any dose of avelumab and have at least one valid ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants
  Participants With Anti-drug Antibodies | 1 | 0
  Participants With Neutralizing Antibodies | 1 | 0

15. Secondary Outcome: Number of Participants With Positive Tumor Programmed Death Ligand 1 (PD-L1) Expression
Description: Number of participants with positive tumor programmed death ligand 1 (PDL-1) with cut off >=1%, >= 5%, >=25%, >=50% and >=80% expression were reported.
Time Frame: Baseline up to end of treatment visit (27.5 weeks)
Population: Biomarker Analysis Set included all participants who received any dose of avelumab and who have provided at least one blood, serum, plasma, or tumor sample for biomarker assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants
  PD-L1 expression at cut-off (>=)1% | 0 | 5
  PD-L1 expression at cut-off of >=5% | 0 | 4
  PD-L1 expression at cut-off of >=25% | 0 | 3
  PD-L1 expression at cut-off of >=50% | 0 | 2
  PD-L1 expression at cut-off of >=80% | 0 | 2

16. Secondary Outcome: Number of Participants With Substantial, Sustained, or Significant Changes From Baseline for Tumor-Infiltrating T-cell Levels
Description: Number of participants with substantial, sustained, or significant changes from baseline for Tumor-Infiltrating T-cell Levels were reported. Significant clinical deterioration (clinical progression), defined as new symptoms that are deemed by the Investigator to be clinically significant or significant worsening of existing symptoms.
Time Frame: Baseline up to end of treatment visit (27.5 weeks)
Population: Since all evaluable tumor tissue samples were collected at baseline and no evaluable sample was provided at end of treatment as planned, an analysis of participants with substantial, sustained, or significant changes from baseline for tumor-infiltrating T-cell levels could not be performed.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Participants With Substantial, Sustained, or Significant Changes From Baseline for T-cell Population in Blood
Description: Number of participants with substantial, sustained, or significant changes from baseline for T-cell population in blood were reported. Significant clinical deterioration (clinical progression), defined as new symptoms that are deemed by the Investigator to be clinically significant or significant worsening of existing symptoms.
Time Frame: Baseline up to end of treatment visit (27.5 weeks)
Population: Due to early termination of the study, the data for this outcome measure was not collected.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Participants With Substantial, Sustained, or Significant Changes From Baseline for B-cell and Natural Killer Cell (NK-Cell) in Blood
Description: Number of participants with substantial, sustained, or significant changes from baseline for B-cell and NK-cell in blood were reported. Significant clinical deterioration (clinical progression), defined as new symptoms that are deemed by the Investigator to be clinically significant or significant worsening of existing symptoms.
Time Frame: Baseline up to end of treatment visit (27.5 weeks)
Population: Due to early termination of the study, the data for this outcome measure was not collected.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants With Substantial, Sustained, or Significant Changes From Baseline for Vaccination-Related Antibody Concentrations
Description: Samples for the testing of vaccination-related antibody concentrations for diphtheria, tetanus, and pneumococcal conjugate (PCV-7) were collected. Significant clinical deterioration (clinical progression), defined as new symptoms that are deemed by the Investigator to be clinically significant or significant worsening of existing symptoms.
Time Frame: Baseline up to end of treatment visit (27.5 weeks)
Population: Due to early termination of the study, the data for this outcome measure was not collected.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs That Resulted in Treatment Discontinuation
Description: Vital signs included: Body temperature, Heart Rate, Blood pressure and respiratory rate. Vital signs were measured in semi-supine position after 5 minutes rest for the participants.
Time Frame: Baseline up to 1182 days
Population: The safety analysis set included all participants who received any dose of avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
Number analyzed (Participants) | 6 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 1182 days
Description: The Adverse Events reported under Serious AEs are the AEs (including non-serious as well as serious AEs) as no separate non-serious AEs were generated as per planned analysis.
Arm/Group | Avelumab 10 Miligram Per Kilogram (mg/kg) | Avelumab 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 6/6 | 12/15
Serious Adverse Events (participants affected / at risk) | 6/6 | 15/15
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab 10 Miligram Per Kilogram (mg/kg) (N=6) | Avelumab 20 mg/kg (N=15)
Thrombocytopaenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 2 | 10
Influenza like illness (General disorders) | 0 | 2
Pyrexia (General disorders) | 4 | 13
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Headache (Nervous system disorders) | 0 | 6
Intracranial pressure increased (Nervous system disorders) | 0 | 2
Pelvic venous thrombosis (Vascular disorders) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 5
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Diplopia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 5
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 6
Stomatitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 6
Asthenia (General disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 3
Fatigue (General disorders) | 0 | 6
Gait disturbance (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pyuria (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 3
Alanine aminotransferase increased (Investigations) | 2 | 0
Amylase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 2
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Device occlusion (Product Issues) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Renal tubular disorder (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 3
Lymphoedema (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was planned to be conducted in 2 parts: the dose-finding part (Phase I) and the tumor-specified expansion part (Phase II). However, Phase II was cancelled due to limited clinical benefit of PD-L1 monotherapy in pediatric participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/25/NCT03451825/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT03451825/SAP_001.pdf